CLINICAL TRIAL: NCT06789692
Title: Reduce Tobacco Use in People Living With HIV in Switzerland: A Pragmatic Randomized Trial Within the Swiss HIV Cohort Study
Brief Title: Reduce Tobacco Use in People Living With HIV in Switzerland
Acronym: RETUNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Novartis Foundation for Medical-Biological Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-02417; ub25Briel
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: HIV; Smoking
Keywords: tobacco smoking; e-cigarettes; tobacco-free nicotine pouches; Trials within Cohorts (TwiCs)
MeSH Terms: conditions — Smoking; Tobacco Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial using the Trials within Cohorts (TwiCs) design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoking substitution menu (Experimental): Offer of preference-based smoking substitution menu, consisting of e-cigarettes or nicotine pouches or nicotine patches in addition to standard of care.
  Interventions: Other: tobacco smoking substitution products
- Standard of care group (No Intervention): Standard smoking cessation counselling according to routine care in the SHCS.

INTERVENTIONS:
Other: tobacco smoking substitution products — Offer of preference-based smoking substitution menu, consisting of e-cigarettes or nicotine pouches or nicotine patches in addition to standard of care. This menu will be offered by the treating physician during the routine cohort visit and the participant can choose one product to test as an alternative to tobacco smoking. The products will be handed out directly after the consultation and are provided free of charge for 6 months.
  Arms: Smoking substitution menu

SUMMARY:
The purpose of this trial is to test the effectiveness of offering a menu of different tobacco smoking substitutional products (e-cigarettes, nicotine pouches, nicotine patches in addition to usual of care) for smokers in the SHCS (Swiss HIV Cohort Study) in achieving self-reported 7-day tobacco cigarette abstinence at 6 months.

DETAILED DESCRIPTION:
Due to highly effective antiretroviral therapy, people living with HIV (PLWH) in Switzerland have a close-to-normal life expectancy. Among PLWH, there has been a shift of focus from HIV-related health issues to non communicable diseases, especially cardiovascular diseases (CVDs) and cancer. Smoking, a prominent risk factor for both diseases, takes a key role in view of the high number of smokers among PLWH.

New approaches to smoking cessation focus on harm reduction by substituting tobacco cigarettes by less harmful alternatives. Conventional nicotine replacement therapy like nicotine patches is well established and effective against withdrawal symptoms after quitting. However, these products are exceptionally expensive and the missing "nicotine hit" often limits therapy adherence. The long-term abstinence rate remains low. Electronic cigarettes (e-cigarettes) and nicotine pouches as alternative nicotine replacement therapies have the potential to overcome these problems and are accessible.

E-cigarettes play a growing role in smoking cessation therapy. Evidence from randomized trials shows superiority over conventional nicotine replacement therapies, which is probably based on the better imitation of the smoking experience. Although e-cigarettes are not without concerns, there is consensus that they are significantly less harmful than tobacco cigarettes.

Tobacco-free nicotine pouches, delivering nicotine through oral mucosa, are a relatively novel option for nicotine substitution. Similar to e-cigarettes, nicotine pouches are relatively affordable and can address the limitation of poor imitation of the "nicotine hit" seen with traditional nicotine replacement therapy. To the best of our knowledge, no trials have investigated the potential of nicotine pouches for smoking cessation so far.

With this trial, the investigators also want to address frequent shortcomings of smoking cessation trials, such as restrictive inclusion criteria and highly controlled interventions, by RETUNE Version 1.1, January 06, 2025 10/45 offering a menu of different tobacco smoking substitutional products (e-cigarettes or nicotine pouches or nicotine patches) and by using a novel pragmatic trial design, the Trials within Cohorts (TwiCs) design. The investigators plan to recruit tobacco smokers in the Swiss HIV Cohort Study (SHCS), regardless of their willingness to quit. This so called "opt-out-approach" has been suggested as a new promising approach for smoking cessation trials to increase generalizability of the results. The TwiCs design optimally allows to implement and evaluate the "opt-out" approach embedded in the SHCS.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for the data collection and participation in the SHCS (Cohort consent).
* Signed informed consent to be randomized to future interventions (Randomization consent).
* Age 18 years or older.
* Smoked one or more tobacco cigarettes per day (smoking status = yes) at the time of enrolment.

Exclusion Criteria:

* Currently using e-cigarettes or nicotine pouches or nicotine patches.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 972 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Tobacco smoking status (yes/no) | at 6 month visit
  Measured as self-reported abstinence in the last 7 day at 6-month visit

SECONDARY OUTCOMES:
Tobacco smoking status (yes/no) | at 12 month visit, 24-month visit
  Measured as self-reported abstinence in the last 7 day at 12-month visit and at 24-month visit
Mean change in number of tobacco-based cigarettes smoked per day | at 6 month visit, at 12 month visit, at 24 month visit
  Number will be self reported by participant
Mean Change in Cholesterol (mmol/l) | at 6 month visit, at 12 month visit, at 24 month visit
  High Density Lipoprotein (HDL) and Low Density Lipoprotein (LDL) Cholesterol in blood samples will be measured
Mean change in blood pressure (mmHg) | at 6 month visit, at 12 month visit, at 24 month visit
  systolic and diastolic blood pressure will be measured.
Mean change in body weight (kg) | at 6 month visit, at 12 month visit, at 24 month visit
  Mean change in body weight from baseline to 6,12 and 24 months.
Mean change in SCORE2-risk prediction algorithm | at 6 month visit, at 12 month visit, at 24 month visit
  SCORE2: Algorithm to Predict Cardiovascular Disease Risk in Europe Linear regression model adjusted for the variables used in the minimization (region [French vs. German speaking part of Switzerland], men having sex with men [yes/no], current drug user [yes/no], number of cigarettes per day) and will be reported as an adjusted odds ratio with 95% confidence interval.
Number of cardiovascular events | at 6 month visit, at 12 month visit, at 24 month visit
  Occurrence of cardiovascular events (myocardial infarction, coronary angioplasty/stenting, coronary artery by-pass grafting, carotid endarterectomy, stroke, deep vein thrombosis, pulmonary embolism, heart transplantation) and all-cause death
Serious Adverse events | at 6 month visit, at 12 month visit, at 24 month visit
  This endpoint will be presented descriptively.
Self reported use of any nicotine containing product other than tobacco cigarettes (yes/no) | at 6 month visit, at 12 month visit, at 24 month visit
Self reported use of e-cigarettes (yes/no) or nicotine pouches (yes/no) or nicotine patches (yes/no) | at 6 month visit, at 12 month visit, at 24 month visit
Self reported use of any nicotine containing product (yes/no) | at 6 month visit, at 12 month visit, at 24 month visit

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Briel, Prof., Principal Investigator — University Hospital, Basel, Switzerland; Alain Amstutz, Dr., Principal Investigator — University Hospital, Basel, Switzerland; Christof Schönenberger, Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (7):
- Switzerland (7):
  - Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - University Hospital Lausanne, Lausanne, Canton of Vaud
  - Cantonal Hospital Aarau, Aarau
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - University Hospital Geneva, Geneva
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (1):
  • Study Protocol (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT06789692/Prot_001.pdf